CLINICAL TRIAL: NCT03779620
Title: Prospective, Controlled, Single-arm Clinical Investigation for the Treatment of Subjects With Severe Symptomatic Aortic Valve Stenosis Using Valvosoft® Pulsed Cavitational Ultrasound Therapy (PCUT) - First-In-Man
Brief Title: Valvosoft First-In-Man Study in Severe Symptomatic Aortic Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiawave SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CW19-01
Record Dates: First submitted 2018-11-12; First posted 2018-12-19 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Aortic Valve Stenosis
Keywords: symptomatic; aortic valve; stenosis; ultrasound; non-invasive
MeSH Terms: conditions — Aortic Valve Stenosis; Constriction, Pathologic

STUDY DESIGN:
Intervention Model Description: Ultrasound treatment of calcified aortic valve stenosis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound treatment (Experimental): Ultrasound treatment of patients with symptomatic aortic valve stenosis who are not eligible for valve replacement
  Interventions: Device: Ultrasound treatment of Calcified aortic valve

INTERVENTIONS:
Device: Ultrasound treatment of Calcified aortic valve — Ultrasound treatment of calcified aortic valve causing symptomatic aortic valve stenosis in patients who are not eligible for valve replacement

SUMMARY:
This is a prospective, controlled, single-arm clinical investigation for the treatment of subjects with severe symptomatic aortic valve stenosis using Valvosoft® Pulsed Cavitational Ultrasound Therapy (PCUT) - First-In-man

DETAILED DESCRIPTION:
CARDIAWAVE has developed a new non-invasive, real-time image-guided, therapeutic approach to treat patients suffering from Calcified Aortic Stenosis. CARDIAWAVE's Valvosoft device is a new ultrasound therapy based on a disruptive technology involving delivering an extremely precise and focused ultrasound beam to perform a reparative effect on the aortic valve leaflets, softening the valve's tissues, restoring leaflet mobility, and therefore improving the overall clinical status related to the aortic valve stenosis. This is a FIM study

ELIGIBILITY:
Inclusion Criteria:

1. Subjects suffering from severe symptomatic aortic valve stenosis (including subjects with a bicuspid valve).
2. Patient is not eligible for TAVR/SAVR .
3. Age ≥18 years.
4. Subjects who are willing to provide a written informed consent prior to participating in the study.
5. Subjects who can comply with the study follow up or other study requirements.
6. Subject eligible according to Clinical Review Committee

   -

Exclusion Criteria:

1. Subjects with any electrical device implanted.
2. Subjects with unstable arrhythmia not controlled by medical treatment.
3. Subjects with implanted mechanical valve in any position or bio prosthetic valve in aortic position.
4. Subjects with complex congenital heart disease.
5. Chest deformity.
6. Cardiogenic shock.
7. History of heart transplant.
8. Subjects requiring other cardiac surgery procedures (bypass graft surgery, mitral valve procedure, tricuspid valve procedure) within one month after treatment.
9. Thrombus in heart.
10. Acute myocardial infarction (MI), stroke or transient ischemic attack (TIA) within one month prior to enrolment*.
11. Subjects who are pregnant or nursing.
12. Subjects who are participating in another research study for which the primary endpoint has not been reached.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Safety: Rate of procedure related mortality at 30 days | 30 days post-procedure
  Rate of procedure related mortality at 30 days
Device performance to modify valve structure as measured by echocardiography | Immediately post-procedure
  Ability to modify the Aortic Valve Area (mm2)
Device performance to modify valve structure as measured by echocardiography | Immediately post-procedure
  Ability to modify the Pressure Gradient (mmHg)

SECONDARY OUTCOMES:
All-cause mortality and major adverse events (MAE's) | Up to 24 months
  Rate of all-cause mortality and MAE's peri and postprocedure and at 1, 3, 6, 12 and 24 months post operatively.
Non-disabling stroke | Up to 24 months
  Rate of stroke at 1,3,6, 12 and 24 months
Improvement of clinical status | Up to 24 months
  Improvement of New York Heart Association class (I-IV - stage of severity of heart failure - I=no symptoms, IV= symptoms at rest) at 1,3,6,12, and 24 months.
Number of all Adverse Events (AEs) | Up to 24 months
  Rate of AE's reported at at 1, 3, 6, 12 and 24 months
User handeling of Valvosoft | Immediately post-procedure
  User handling (questionnaire for operator + procedure duration) immediately post-procedure
Improvement of quality of life | upto 24 months
  Improvement of quality of life by means of Kansas City Cardiomyopathy Questionnaire at 1, 3, 6, 12 and 24 months
Long term maintenance of improvement of AVA and PG | upto 24 months
  Long term maintenance of improvement of AVA and PG at 3, 6, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Messas, MD, Principal Investigator — HGEP Paris, France
Locations (2):
- Hôpital Européen Georges Pompidou, Paris, France
- Amphia Hospital, Breda, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Messas E, Ijsselmuiden A, Trifunovic-Zamaklar D, Cholley B, Puymirat E, Halim J, Karan R, van Gameren M, Terzic D, Milicevic V, Tanter M, Pernot M, Goudot G. Treatment of severe symptomatic aortic valve stenosis using non-invasive ultrasound therapy: a cohort study. Lancet. 2023 Dec 16;402(10419):2317-2325. doi: 10.1016/S0140-6736(23)01518-0. Epub 2023 Nov 14. PMID 37972628
- [Derived] Messas E, IJsselmuiden A, Goudot G, Vlieger S, Zarka S, Puymirat E, Cholley B, Spaulding C, Hagege AA, Marijon E, Tanter M, Bertrand B, Remond MC, Penot R, Ren B, den Heijer P, Pernot M, Spaargaren R. Feasibility and Performance of Noninvasive Ultrasound Therapy in Patients With Severe Symptomatic Aortic Valve Stenosis: A First-in-Human Study. Circulation. 2021 Mar 2;143(9):968-970. doi: 10.1161/CIRCULATIONAHA.120.050672. Epub 2021 Jan 25. No abstract available. PMID 33486971